CLINICAL TRIAL: NCT07151040
Title: A First-in-human, Phase 1/2, Multicenter, Open-label, Dose Escalation, Confirmation and Expansion Study to Evaluate the Safety, Pharmacokinetics and Antitumor Activity of TH9619 in Subjects With Advanced Solid Tumors
Brief Title: Phase 1/2 Study to Evaluate TH9619 in the Treatment of Advanced Solid Tumors
Acronym: ODIN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: One-carbon Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH9619-0101; 2024-519639-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-13; First posted 2025-09-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Colorectal Cancer (CRC); Squamous Cell Carcinoma of Head and Neck; Non-Small Cell Lung Cancer (NSCLC); Gastrooesophageal Junction Cancer; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm dose (Experimental): Phase 1a (escalation) Single arm dose escalation of TH9619 as monotherapy. Phase 1b (expansion) Single arm dose expansion of TH9619 as monotherapy in selected tumor types.
  Interventions: Drug: TH9619

INTERVENTIONS:
Drug: TH9619 — Phase 1a - DOSE ESCALATION
  Description:
  Single arm dose escalation of TH9619 as monotherapy.
  Phase 1b - DOSE EXPANSION
  Description:
  Single arm dose expansion of TH9619 as monotherapy in selected tumor types. The objectives and endpoints for the expansion cohort(s) will be defined in a protocol amendment, once data from Phase 1a are available.

SUMMARY:
This is a first in human, multi-center, open-label, dosage escalation study to determine the recommended dose range of TH9619 in subjects with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent
* Histopathologically confirmed advanced cancer (colorectal cancer, head and neck squamous cell cancer, non-small cell lung cancer and gastric cancer (including gastroesophageal junction cancer))
* Prior treatment with at least one line of cytotoxic systemic therapy for metastatic/unresectable cancer
* Adult patients (≥18 years of age)
* Must be willing to comply with study procedures

Exclusion Criteria:

• History or presence of any clinically significant disorders as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs) | From the start of Cycle 1 Day 1, through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of severe treatment-emergent adverse events (TEAEs) per Common Terminology for Adverse Events (CTCAE) V5.0 grading | From the start of Cycle 1 Day 1, through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of treatment-emergent adverse events (TEAEs) related to treatment, as assessed by the Investigator | From the start of Cycle 1 Day 1, through the 28-day study treatment cycles and follow-up, up to 2 years.
Frequency of serious adverse events (SAEs) | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of serious adverse events (SAEs) per the seriousness criteria defined in the protocol. | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of serious adverse events (SAEs) related to treatment, as assessed by the Investigator | From the start of Cycle 1 Day 1, through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of out of range clinical laboratory tests (as defined by the clinic) assessed as clinically significant by the Investigator | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of findings on vital signs parameters assessed as clinically significant by the Investigator | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of findings on ECHO/ECG assessed as clinically significant by the Investigator | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of findings during physical examinations assessed as clinically significant by the Investigator | From the screening visit (maximum 28 days from Cycle 1 Day 1), through the 28-day study treatment cycles and follow-up, up to 2 years.
Incidence of treatment emergent adverse events (TEAEs) leading to dose interruptions/reductions and/or discontinuation of treatment | From the start of Cycle 1 Day 1, through the 28-day study treatment cycles and follow-up, up to 2 years.

CONTACTS AND LOCATIONS:
Locations (4):
- Institut Gustave Roussy, Villejuif, France
- Spain (2):
  - Vall D Hebron Institute Of Oncology, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
- Newcastle University, Newcastle upon Tyne, United Kingdom